CLINICAL TRIAL: NCT06780319
Title: Digital Rehabilitation After Hip Arthroplasty: a Randomized Controlled Trial
Acronym: Digihip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Sport, Bordeaux Mérignac (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-17-SBM
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hip Arthroplasty, Total
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard rehabilitation (Active Comparator)
  Interventions: Procedure: Standard rehabilitation
- Tele-rehabilitation (Experimental)
  Interventions: Procedure: Tele-rehabilitation

INTERVENTIONS:
Procedure: Standard rehabilitation — rehabilitation with a private physiotherapist. Patients usually undergo 15 rehabilitation sessions, in line with HAS recommendations; the number of sessions can go up to 25, depending on the patient's profile and needs.
  Arms: standard rehabilitation
Procedure: Tele-rehabilitation — Tele-education is a digital home-based intervention involving exercises and education. Patients are monitored remotely by a physiotherapist via a secure messaging system. The system consists of a mobile application for the patient and a web portal enabling the physiotherapist to review patient data (physical activity, pain levels, medication use, exercise adherence, patient-reported results, images, videos) on a daily basis and tailor the protocol accordingly.
  Arms: Tele-rehabilitation

SUMMARY:
The study aims to compare the effectiveness of tele-rehabilitation versus no physical therapy after total hip arthroplasty (THA) in improving patient-reported outcomes and functional recovery. THR is a common surgical procedure to relieve pain and improve function in patients with a variety of hip conditions. Traditional physical therapy is a standard component of the post-operative care pathway for PTH patients, but can be hampered by logistical obstacles. Tele-rehabilitation is emerging as a promising alternative, offering the potential to overcome these barriers and improve access to care. The study uses a prospective monocentric design with two arms and a follow-up time of 6 months. The primary objective is assessed using the Timed up and go Test (TUG), while secondary objectives include patient-reported outcome measures, patient satisfaction, healthcare utilization, and return to physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Have an email address and a smartphone
* Patient speaking and writing French
* Patient covered by a social security scheme

Exclusion Criteria:

* Hip revision surgery, significant comorbidities (Parkinson's disease, multiple sclerosis, stroke) or psychiatric disorders (substance use) that could interfere with rehabilitation
* Patients with disorders that make it difficult for them to express their feelings
* Pregnant or breast-feeding patients
* Patient under protective supervision
* Patient not covered by a social security scheme

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Time Up and Go test | 6 weeks and 6 months after surgery
  The TUG is a clinical test used to assess patients' mobility and risk of falling. It measures the time required for a person to stand up from a chair, walk a short distance, turn around, return to the chair and sit down.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport, Mérignac, France

IPD SHARING:
Plan to Share IPD: No